CLINICAL TRIAL: NCT05997940
Title: Evaluation Of The Postoperative Analgesic Effectiveness Of The Pericapsular Nerve Group Block Performed Before Spinal Anesthesia In Hip Surgery
Brief Title: Effectiveness Of The Pericapsular Nerve Group (PENG) Block In Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Mustafa Ogurlu, Professor Doctor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022/03
Record Dates: First submitted 2023-07-11; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: PENG Block
Keywords: Pericapsular nerve group (PENG) block; Postoperative analgesia; Hip Surgery; Regional anesthesia; Spinal anesthesia
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG (Active Comparator): PENG block performed before spinal anesthesia
  Interventions: Drug: PENG block
- Control (No Intervention)

INTERVENTIONS:
Drug: PENG block — The PENG block was performed with the patient in the supine position at preoperative waiting room. A curvilinear low-frequency ultrasound probe (2-5 MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22 gauge, 100 mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution was injected in 5 mL increments while observing for adequate fluid spread in this plane for a total volume of 20 mL
  Arms: PENG

SUMMARY:
The target population of hip surgery is usually the elderly patients with systemic comorbidity. Especially hip fractures are common in society and cause high morbidity and mortality for geriatric patients . Pain felt before and during surgery can cause metabolic and endocrine changes in the body, leading to sleep disorders, depression, delirium, dementia and persistent chronic pain. With effective postoperative analgesia, it is possible to reduce postoperative complications and mortality and accelerate post-surgical recovery. Pharmacological methods such as opioids and NSAIDs used for this may cause further deterioration and other side effects in geriatric patients with reduced renal and hepatic function, thus delaying post-surgical recovery and thus discharge. In order to avoid these side effects, regional anesthesia techniques can be preferred.

Regional anesthesia techniques are among the most effective methods of postoperative analgesia. Peripheral nerve blocks are also one of the regional anesthesia methods. Peripheral nerve blocks; They are the most ideal postoperative analgesia methods because they provide effective analgesia, reduce the need for opioids and consequently their side effects, are effective in the treatment of dynamic pain and facilitate recovery.

Patients undergoing hip surgery have very severe pain and need additional postoperative analgesics. Mobilization of patients is delayed due to pain . Depending on this , thromboembolism , deep vein The risk of nosocomial infection increases due to thrombosis , wound infection and increased length of stay.

Alleviating the pain around the hip joint capsule is an effective analgesia method in hip surgeries. The anterior capsule of the hip joint is innervated by the femoral , obturator , and accessory obturator nerves . Pericapsular nerve group (PENG) block also targets these nerves. Many studies have shown that PENG block provides adequate analgesia for more than 24 hours postoperatively. PENG block is a method that is frequently used in the world and in our clinic and has a low complication rate.

In this study, the investigators aimed to show that pericapsular nerve group block performed before spinal anesthesia in hip surgeries reduces postoperative pain and decreases total opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients with written informed consent
* Patients over 18 years old
* Patients with ASA score I-II-III
* Patients performed spinal anesthesia for surgery

Exclusion Criteria:

* Patients without written informed consent
* Patients with ASA score IV and above
* Patients who cannot be communicated
* Patients with infection at the block site
* Patients with coagulation disorders
* Patients not suitable for spinal anesthesia
* Patients with liver and kidney failure
* Patients who are allergic to the drugs used
* Patients with major complications during the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Preoperative
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | During the spinal anesthesia
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Postoperative 0. hour
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Postoperative 1. hour
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Postoperative 6. hour
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Postoperative 12. hour
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).
Numeric Rating Scale (NRS) for postoperative analgesic efficacy | Postoperative 24. hour
  NRS is a one-dimensional scale used to measure pain intensity. The patient is asked to select the number that best describes the level of pain as 0 = no pain and 10 = worst pain (unbearable).

SECONDARY OUTCOMES:
Amounts of postoperative analgesic consumption | Postoperative 24 hours
  Postoperative analgesic consumption amounts will be compared between the patients performed PENG block and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Turkey (Türkiye)